CLINICAL TRIAL: NCT02828826
Title: Impact of Telephone Coaching on Physical Performance in a Physical Exercise Maintenance Program for Fallers Elderly Patients Living at Home
Acronym: STEP-PA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion deficiency
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC16_0030
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2018-03

CONDITIONS: Fall

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telephone coaching (Experimental): Patients randomized to the experimental group will benefit from the telephone coaching , with 5 phone calls programmed by the physiotherapist according to the most convenient times for the patient, due to appointments per month.
  The telephone coaching conducted by the physiotherapist with patients is to assess the number of exercises performed, the number of falls may have occurred, assess the fear of falling and overall assessment of the patient's general condition and a self-assessment of their physical ability (one leg balance, fear of falling, FTSST). With this information, the therapist may encourage patients to practice more diligently exercises can even strengthen the practice of some based on its evaluation.
  Data from the telephone coaching will be recorded in the eCRF.
  Interventions: Other: telephone coaching
- Without telephone coaching (No Intervention)

INTERVENTIONS:
Other: telephone coaching
  Arms: telephone coaching

SUMMARY:
At home, maintenance, physical performance declines more or less rapidly from 6 weeks depending advancing age and duration of the training period . It is feared that the advice or prescription of regular physical maintenance at the exit of the service, has only adherence to the 50% like the medication prescribed. A US study of 2000 on the observance of healthy living recommendations, despite the many messages promoting physical activity, shows that only 24% of Americans aged 65 to 74 were taking physical activity regular. There are no French-date data.

If physical maintenance is routinely recommended for the elderly living at home, so the way to encourage these people to practice more often possible these recommendations remains therefore a problem of public health.

The recent OSSEBO study (intervention for the prevention of injurious falls in elderly women: background and design) recalled the interest to propose a program of physical exercise to reduce trauma and falls in the elderly. It also shows the possibility to implement an effective program on a long-term and large scale in France. The study allowed patients to participate in collective sessions of physical exercises, within the framework of an association. Patients were invited to continue their home exercises they had learned.

Also, the investigators hypothesize that the monthly telephone coaching , directed by the physical therapist following a physical fitness exercise program which they have been trained during their hospitalization in SSR , would allow older patients to maintain fallers their physical performance at home for at least 6 months after leaving

DETAILED DESCRIPTION:
Before to the start of the study, physical therapists and CRA (clinical research associate) will be trained in the specifics of this research protocol.

Patients aged 65 and older, with physiotherapy treatment, investigators will be offered to participate in the study.

The physiotherapist of the investigative service will inform the patient of the terms of the study and will give the necessary information on the physical maintenance program, (presenting the program, verification of the correct understanding of the program and it ran properly, recall the entry on a calendar associated to the program booklet whenever the program achieved, advice on the interests of the exercises as many times as possible per week).

If the patient agrees to participate, the physical therapist will give him a copy of the prospectus and gather written consent after a delay of 24 hours.

The patient will receive the booklet detailing the physical exercise program and allowing him to record his achievement of physical exercise and its possible falls.

Following the inclusion of the patient, the physiotherapist will inform the computerized data file and will proceed to randomization via Clinsight® software.

The patient will be informed of the group in which it is randomized (with or without telephone coaching ) .

The patient will receive a summons for assessments to M6 and M12 to be carried on the website of the investigation center . It will be recalled him to bring his book.

Before its release SSR ( M0 ), the patient will benefit included in the initial assessment including a TUG ( Score Time UP and Go), VAS (Visual Analog Scale ) measures the fear of falling , the IADL (INSTRUMENTAL ACTIVITIES OF DAILY LIVING), the FTSST (Five Times Sit to Stand Test) and score the one leg balance test . The running score 4 meters. This initial evaluation will be conducted by the physiotherapist or the CRA by location Patients randomized to the control group will not receive telephone coaching . Patients will only record the achievement of physical exercises and the occurrence of falls in their booklet.

Patients randomized to the experimental group will benefit from the telephone coaching , with 5 phone calls programmed by the physiotherapist according to the most convenient times for the patient, due to appointments per month.

The duration of each telephone coaching is estimated at 20mn . As patients in the control arm , Patients will record their physical exercise sessions and the occurrence of falls in their booklet.

The telephone coaching conducted by the physiotherapist with patients is to assess the number of exercises performed, the number of falls may have occurred, assess the fear of falling and overall assessment of the patient's general condition and a self-assessment of their physical ability (one leg balance, fear of falling, FTSST). With this information, the therapist may encourage patients to practice more diligently exercises can even strengthen the practice of some based on its evaluation.

Data from the telephone coaching will be recorded in the eCRF ( Case Report Form).

A M6, the patients in both study arms will receive an evaluation including a TUG, EVA measures the fear of falling, the IADL, the FTSST, walking speed and score the one leg balance test. The number of re hospitalizations and use of a physiotherapist for motor rehabilitation will also be sought from the patient and her doctor if necessary. This evaluation will be carried out by a TEC, as part of a consultation center investigator.

At the end of the evaluation M6, patients in the experimental arm no longer benefit from telephone coaching. As for patients in the control arm, they will only record their exercise sessions and the occurrence of falls in their booklet.

A final evaluation of patients will be performed at M12 (same as M6) Following the visits and phone calls, the study data will be recorded in the eCRF by the CRA and / or physiotherapist investigators centers.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 65 and over
* Patient having a physiotherapy treatment
* Faller patient ( a fall in the preceding 12 months)
* patient leaving the service to return home or living at home
* Patient with a score ≥ 24/30 in the Mini Mental Status (MMS )
* patient able to get up a seat and walk 6 meters without human assistance (corresponds to test TUG ) patient
* informed of the study has given free and informed consent

Exclusion Criteria:

* Patient under judicial protection , under guardianship
* patient with active disease , with degenerative impact on walking,
* patient unable to use the phone
* patient with visual impairments preventing reading the physical maintenance program
* Refusal of patient participation
* Patient not wishing to stop his liberal physiotherapy care to driving
* Patient included in another interventional research protocol

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Score ̏ Timed Up and Go ( TUG ) at 6 months of SSR output | 6 months
  The test is simple, attainable in 3 minutes in a quiet room with no noise with a standard chair with armrests. A line is marked on the ground at 3m from the chair. The examiner, provides with a stopwatch, should not encourage the patient. The patient performs the test with his shoes and his usual technical assistance. The patient should walk at a comfortable pace and as naturally as possible. The patient will have to stand up, turn around and return to the line sit.
  The test is performed 2 times: once to verify that the patient understands the instructions, then again timed.
  Reproducing the test has a degree of correlation between r = 0.92 and 0.99. There is excellent agreement between the various evaluators (0.93 to 0.99 correlation coefficient) (49).
  The TUG shows good diagnostic validity with a sensitivity and a specificity of 87% for the fall prediction .

SECONDARY OUTCOMES:
Score ̏ Timed Up and Go ( TUG ) at 12 months of SSR output | 12 months
number of falls reported by the patient | 6 months
number of falls reported by the patient | 12 months
fear of falling | 6 months
  assessing the fear of falling on a visual analogue scale
fear of falling | 12 months
  assessing the fear of falling on a visual analogue scale
score of autonomy with the IADL (Instrumental Activities of Daily Living ) | 6 months
score of autonomy with the IADL (Instrumental Activities of Daily Living ) | 12 months
score of FTSST (Five Timed Sit to Stand Test) | 6 months
  performance of the lower limbs
score of FTSST (Five Timed Sit to Stand Test) | 12 months
  performance of the lower limbs
number of re hospitalization for fall | 6 months
number of re hospitalization for fall | 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Ch Cholet, Cholet
  - Centre hospitalier départemental Vendée, La Roche-sur-Yon
  - SSR du Château de Marlonges Groupe Hospitalier La Rochelle, La Rochelle
  - CH Emile Roux, Le Puy-en-Velay
  - CHD Vendée Montaingu, Montaigu
  - Cabinet Liberal Martin, Nantes
  - CHU de Nantes, Nantes
  - Centre Le Bodio, Pontchâteau
  - MSP Pôle Santé du Marais, Saint-Gervais
  - CH Saint-Nazaire, Saint-Nazaire

REFERENCES:
- [Derived] Rince G, Volteau C, Fortin J, Couturier CC, Rulleau T. Impact of telephone coaching supporting a physical maintenance exercise programme for older adults at risk of falls: a randomised controlled trial. BMC Geriatr. 2024 Oct 26;24(1):879. doi: 10.1186/s12877-024-05488-y. PMID 39462354